CLINICAL TRIAL: NCT01897558
Title: Effect of Passive Versus Active Fixation Leads on the Magnitude of Troponin Release After Pacemaker Implantation (PACMAN Trial)
Brief Title: Myocardial Micro-damage in Relation to Active and Passive Fixation Pacemaker Electrodes
Acronym: PACMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GER-EP-012
Record Dates: First submitted 2013-05-02; First posted 2013-07-12 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Bradyarrhythmia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ventricular pacemaker electrode (Active Comparator): receives an active fixation ventricular pacemaker electrode
  Interventions: Device: Pacemaker implantation
- Passive fixation ventricular pacemaker electrode (Active Comparator): receives a passive fixation ventricular pacemaker electrode
  Interventions: Device: Pacemaker implantation

INTERVENTIONS:
Device: Pacemaker implantation

SUMMARY:
Pacemaker electrodes are either equipped with tines (passive fixation) or with a screw (active fixation) for initial fixation in the patient´s heart. Both types of electrodes provide similar results in a long-term follow-up and the use of one or the other electrode type in many instances is mainly based on the implanter´s preference. The PACMAN-trial investigates whether the two lead types are associated with different amounts of myocardial micro-damage during implantation.

ELIGIBILITY:
Inclusion Criteria:

* de-novo implantation of a pacemaker system

Exclusion Criteria:

* AAI pacing or cardiac resynchronization therapy
* ICD indication
* temporary pacing
* lead revision
* right ventricular pacing aimed from alternative pacing sites (other than the apex)
* lead revision
* severe tricuspid valve regurgitation
* previous myocardial infarction, coronary intervention, stroke, cardioversion or ablation in the presence of elevated troponin levels
* dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
high-sensitive Troponin T | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (5):
- University Hospital Dubrava, Zagreb, Croatia
- Germany (3):
  - Klinikum Kempten, Kempten
  - Krankenhaus Landshut-Achdorf, Landhut
  - Deutsches Herzzentrum München, München
- Kenri Hospital, Mishima, Japan

REFERENCES:
- [Result] Blazek P, Ferri-Certic J, Vrazic H, Lennerz C, Grebmer C, Kaitani K, Karch M, Starcevic B, Semmler V, Kolb C. Pacemaker Implantation Associated Myocardial Micro-Damage: A Randomised Comparison between Active and Passive Fixation Leads. Sci Rep. 2018 Mar 20;8(1):4870. doi: 10.1038/s41598-018-23209-5. PMID 29559697